CLINICAL TRIAL: NCT01463150
Title: Prasugrel 5mg Versus High Dose Clopidogrel in Clopidogrel Resistant Patients Aged ≥75 Years and/or Weighing <60 kg Post Percutaneous Coronary Intervention (PCI)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Patras (Other)
Responsible Party: Principal Investigator, Dimitrios Alexopoulos, Professor, University of Patras
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PATRASCARDIOLOGY-7
Record Dates: First submitted 2011-10-27; First posted 2011-11-01 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-04

CONDITIONS: Platelet Reactivity
Keywords: Platelet reactivity; Clopidogrel; Prasugrel
MeSH Terms: interventions — Clopidogrel; Prasugrel Hydrochloride

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clopidogrel (Active Comparator): Clopidogrel 150mg per day for 15 days
  Interventions: Drug: Clopidogrel
- Prasugrel (Experimental): Prasugrel 5mg for 15 days
  Interventions: Drug: Prasugrel

INTERVENTIONS:
Drug: Clopidogrel — Clopidogrel 150mg per day for 15 days
  Arms: Clopidogrel
Drug: Prasugrel — Prasugrel 5mg per day for 15 days
  Arms: Prasugrel

SUMMARY:
The use of dual antiplatelet therapy is considered standard of care in patients post percutaneous coronary intervention (PCI) with stenting. However, a significant proportion of patients is considered clopidogrel resistant and this resistance is shown to be accompanied by future adverse events. The aim of the study is to define in consecutive patients with acute coronary syndrome (ACS) undergoing PCI, those aged>75years and/or weighted<60 Kg with high on-clopidogrel platelet reactivity (Platelet Reactivity Units-PRU≥235) as estimated 24 hours post PCI with the VerifyNow assay. Those patients will be randomized after informed concent in 1:1 fashion to prasugrel 5 mg or clopidogrel 150mg daily. Platelet reactivity will be assessed at day 15 and then treatment crossover will be performed. At day 30 platelet reactivity will be determined as well.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old
2. Patients having PCI with stenting 24 hours prior randomization, meeting the following criteria :

   * Acute coronary syndrome (unstable angina or myocardial infarction)
   * TIMI risk score>2
3. Platelet reactivity in PRU ≥235 24 hours post-PCI
4. Age≥75 years and/or weight<60 Kg

4. Informed consent obtained in writing

Exclusion Criteria:

* A history of bleeding diathesis
* Chronic oral anticoagulation treatment
* Contraindications to antiplatelet therapy
* Known platelet function disorders
* PCI or coronary artery bypass surgery < 3 months
* Unsuccessful PCI (residual stenosis > 30% or flow < Thrombolysis in myocardial infarction flow 3)
* Planned staged PCI in the next 30 days
* Hemodynamic instability
* hemodialysis
* Creatinine clearance <25 ml/min
* inability to give informed consent
* High likelihood of being unavailable for the Day 30
* History of gastrointestinal bleeding, genitourinary bleeding or other site abnormal bleeding within the previous 6 months.
* Other bleeding diathesis, or considered by investigator to be at high risk for bleeding on longterm antiplatelet therapy.
* Any previous history of ischemic stroke, transient ischemic attack, intracranial hemorrhage or disease (neoplasm, arteriovenous malformation, aneurysm).
* Thrombocytopenia (<100.000 / μL) at randomization
* Anaemia (Hct <30%) at randomization
* Polycythaemia (Hct > 52%) at randomization
* Periprocedural IIb/IIIa inhibitor administration

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2011-10; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Platelet reactivity | 15 days
  Platelet reactivity assessed with the VerifyNow assay at the end of each treatment period

SECONDARY OUTCOMES:
Hyporesponsiveness rate (PRU≥235) at the end of the 2 treatment periods | 15 days
  Hyporesponsiveness rate will be assessed 15 days after the onset of each study drug

CONTACTS AND LOCATIONS:
Locations (1):
- Cardiology Department Patras University Hospital, Rio, Achaia, Greece

REFERENCES:
- [Derived] Alexopoulos D, Xanthopoulou I, Plakomyti TE, Theodoropoulos KC, Mavronasiou E, Damelou A, Hahalis G, Davlouros P. Pharmacodynamic effect of prasugrel 5 mg vs clopidogrel 150 mg in elderly patients with high on-clopidogrel platelet reactivity. Am Heart J. 2013 Jan;165(1):73-9. doi: 10.1016/j.ahj.2012.10.008. Epub 2012 Nov 14. PMID 23237136